CLINICAL TRIAL: NCT02085213
Title: GOT-IT Trial: A Pragmatic Group Sequential Placebo Controlled Randomised Trial to Determine the Effectiveness of Glyceryl Trinitrate for Retained Placenta.
Brief Title: GOT-IT Trial: Glyceryl Trinitrate for Retained Placenta
Acronym: GOT-IT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Aberdeen (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HTA 12/29/01; 2013-003810-42 (EudraCT Number); 12/29/01 (Other Grant/Funding Number: NIHR HTA Programme); 13/NE/0339 (Other: REC Approval)
Record Dates: First submitted 2014-03-04; First posted 2014-03-12 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Placenta, Retained
Keywords: Retained placenta; Manual Removal of Placenta; Glyceryl Trinitrate
MeSH Terms: conditions — Placenta, Retained | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glyceryl Trinitrate (Experimental): Nitrolingual Pump Spray [Coro-Nitro] A liquid within non-pressurised, red plastic-coated glass bottle fitted with a pump capable of delivering a metered dose containing 400μg of glyceryl trinitrate.
  Excipients: The formulation contains fractionated coconut oil, absolute ethanol, medium chain partial glycerides and peppermint oil.
  The treatment will be self administered (2 puffs) as a single intervention. No second intervention will be given.
  Interventions: Drug: Glyceryl Trinitrate
- Placebo (Placebo Comparator): Matched placebo formulation (except for active ingredient of Glyceryl Trinitrate) with matched packaging and labelling.
  Interventions: Drug: Matched Placebo

INTERVENTIONS:
Drug: Glyceryl Trinitrate
  Other Names: GTN
  Arms: Glyceryl Trinitrate
Drug: Matched Placebo — Matched placebo
  Other Names: Dummy treatment
  Arms: Placebo

SUMMARY:
A retained placenta (RP) is a complication after a normal birth, which affects nearly 11,000 women in the UK per year. This is where the placenta is not delivered spontaneously after giving birth. It is a major cause of postpartum haemorrhage (major loss of blood) which can lead to the death of the mother. The recommended treatment for RP is a surgical procedure - manual removal of placenta (MROP). This is a painful and unpleasant intervention for the women, involving additional hospital stay, and is an expensive outcome for the NHS. It is widely recognised that non-surgical management options for RP are limited and it has been recommended that research is needed into new medical treatments for RP. New effective treatments for RP would dramatically reduce the number of women requiring MROP with the operation being restricted to the small minority of women with particularly stuck placentae. The reduction in operative interventions would have cost benefits for the NHS and also for women in terms of increased satisfaction, less separation of mother and baby immediately after birth, and reduced morbidity.

This study will try to prove the clinical and cost effectiveness of a known treatment for angina, Glyceryl trinitrate (GTN) used to treat RP. The investigators will compare GTN against a placebo (dummy treatment) in a randomised controlled blinded trial (GOT-IT).

The GOT-IT Trial will be conducted in two phases. The first phase will involve an internal pilot study where the aim will be to test out and refine trial procedures in a small number of hospital sites. The second phase will be the main trial where recruitment will be extended to a larger number of hospitals in order to determine clinical and cost effectiveness.

DETAILED DESCRIPTION:
Although a growing body of evidence supports a use for GTN for treatment of RP, much of this evidence is based on anecdotal case-reports or clinical "trials" which are non-randomised, do not include a placebo arm and are underpowered. Further, in the context of constrained maternity resources in a publicly funded health system, it is important to quantify the costs associated with the use of GTN (including any subsequent monitoring costs and costs associated with complications) in relation to its effectiveness and any subsequent cost savings it may deliver over standard practice. There is therefore an urgent need for a pragmatic clinical trial of GTN for RP to determine whether GTN is efficacious, safe, acceptable and cost-effective as a treatment for RP before a treatment which may (or may not) work is embedded within routine clinical practice. Our proposed randomised placebo controlled double blind pragmatic UK wide GOT-IT trial RCT (with internal pilot study) will definitively determine whether sublingual GTN is (or is not) clinically and cost effective for management of RP.

ELIGIBILITY:
Inclusion Criteria:

* Women with retained placenta.
* Women aged 16 or over.
* Women with vaginal delivery (including women with a previous caesarean section).
* Haemodynamically stable (systolic blood pressure more than 100mg Hg and pulse less than 110 beats per min).
* > 14 weeks gestation.

Exclusion Criteria:

* Unable to give informed consent.
* Suspected placenta accreta/increta/percreta.
* Multiple pregnancy.
* Women having an instrumental vaginal delivery in theatre
* Allergy or hypersensitivity to nitrates or any other constituent of the formulation.
* Taken alcohol in the last 24 hours.
* Concomitant use with phosphodiesterase inhibitors (such as sildenafil, tadalafil, or vardenafil).
* Contra-indication due to one of the following: Severe anaemia, constrictive pericarditis, extreme bradycardia, incipient glaucoma, Glucose-6- phosphatedehydrogenase-deficiency, cerebral haemorrhage and brain trauma, aortic and / or mitral stenosis and angina caused by hypertrophic obstructive cardiomyopathy. Circulatory collapse, cardiogenic shock and toxic pulmonary oedema.
* Currently participating in another CTIMP.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1107 (Actual)
Dates: Start 2014-09; Primary Completion 2017-07-26 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Need for Manual Removal of Placenta | From time of randomisation up to 15-minutes post administration of study treatment
  Defined as the placenta remaining undelivered 15 minutes post study treatment and/or being required within 15 minutes of treatment due to safety concerns.

SECONDARY OUTCOMES:
Fall in haemoglobin | First postnatal day (approximately 24 hours since the birth).
  Fall in haemoglobin of more than 15% between recruitment and the first postnatal day.
Time from randomisation to delivery of placenta. | From time of randomisation and administration of the study treatment to delivery of placenta (up to approximately 2 hours).
  The time from when the study drug is administered until the placenta is delivered.
Need for earlier than planned MROP on the basis of the clinical condition. | From time of randomisation and administration of the study treatment to delivery of placenta (up to approximately 2 hours).
  This will measure how many women required to go to theatre as an emergency before the 15 minute trial has been completed.
Systolic and diastolic blood pressure. | Study treatment to 15 minutes postadministration.
  Fall in systolic or diastolic blood pressure of more than 15mmHg and/or increase in pulse of more than 20 beats/minute between baseline and 5 and 15 minutes postadministration of active/placebo treatment.
Need for blood transfusion | From the time of delivery of the placenta to time of discharge from hospital (up to 7 days).
  How many women will be required to have a blood transfusion between time of delivery and hospital discharge.
Need for general anaesthesia | From time of randomisation and administration of the study treatment to delivery of placenta (up to approximately 2 hours).
  Will measure how many women required a general anaesthetic from when the study drug was administered until the placenta was delivered.
Maternal Pyrexia | Within 72 hours of delivery or discharge from hospital if discharge occurs sooner
  One or more temperature reading of more than 38°C.
Sustained uterine relaxation. | Within 24 hours of the time of delivery of the placenta.
  Sustained uterine relaxation after removal of placenta requiring uterotonics.
Mean costs for each treatment allocation group | 6 weeks.
  The mean costs will be summarised by treatment allocation group, and the incremental cost (cost saving) associated with the use of GTN will be estimated using an appropriately specified general linear model. The cost data will be presented alongside the primary and secondary outcome data in a cost-consequence balance sheet, indicating which strategy each outcome favours.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona C Denison, Dr, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Derived] Denison FC, Carruthers KF, Hudson J, McPherson G, Chua GN, Peace M, Brewin J, Hallowell N, Scotland G, Lawton J, Norrie J, Norman JE; GOT-IT investigator team. Nitroglycerin for treatment of retained placenta: A randomised, placebo-controlled, multicentre, double-blind trial in the UK. PLoS Med. 2019 Dec 30;16(12):e1003001. doi: 10.1371/journal.pmed.1003001. eCollection 2019 Dec. PMID 31887169